CLINICAL TRIAL: NCT05867927
Title: GENERATE - Next GENERATion of GynEcological Surgery - Robotic Assisted Surgery in Gynecological Indications - A Prospective, Non-interventional, Multi-center, Post Market Clinical Study
Brief Title: GENERATE - Next GENERATion of GynEcological Surgery - Robotic Assisted Surgery in Gynecological Indications
Acronym: GENERATE
Status: Recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 114363C
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: GYN Disorders
MeSH Terms: conditions — Genital Diseases, Female | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- da Vinci Patients: Consecutive enrollment of patients with indications of interest and having a da Vinci robotic-assisted surgery
  Interventions: Device: Robotic-assisted surgery (da Vinci)
- Epidemiological Data Audit: Extended data collection on patients with indications of interest, eligible for a robotic-assisted surgery, but treatment choice was not a da Vinci surgery
  Interventions: Device: Non-da Vinci Surgery

INTERVENTIONS:
Device: Robotic-assisted surgery (da Vinci) — Robotic-assisted surgery (da Vinci)
  Groups: da Vinci Patients
Device: Non-da Vinci Surgery — Non-da Vinci Surgery
  Groups: Epidemiological Data Audit

SUMMARY:
GENERATE - Next GENERATion of GynEcological Surgery - Robotic Assisted Surgery in Gynecological Indications

Generate real-world evidence in the use of the da Vinci Surgical Systems for gynecological indications within the German health care system.

DETAILED DESCRIPTION:
A prospective, non-interventional, multi-center, post market clinical study.

ELIGIBILITY:
Key Inclusion Criteria:

* Woman with 18 years of age or older
* Patient is willing to participate and to comply with the study procedures as demonstrated by signing the informed consent
* Patient is a candidate for a gynecological procedure to be performed with the Intuitive Surgical System

Key Exclusion Criteria:

* Life expectancy of less than 1 year
* Pregnancy, or positive pregnancy test for women prior to menopause or breastfeeding women
* Current participation in a clinical study, if not pre-approved by Intuitive
* Individuals who are unable to fully understand all aspects of the study that are relevant to the decision to participate (mentally or verbally), or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gynecological disease that may be treated by surgical intervention.
Sampling Method: Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of complications related to the surgery up to 30 days | 30 days
  Describe the number of complications related to the surgery up to 30 days; adverse events as documented during the first 30 days will be classified as four different levels of causality to the surgery (not related, possible, probable and causal relationship). Descriptive analysis will be performed.
Describe the number of patient-reported outcomes up to 12 months | 12 months
  Describe the patient-reported outcomes up to 12 months; descriptive analysis will be performed on the data directly reported via the patients (patient questionnaires); information included are number of complications, re-hospitalizations, re-operations, disease recurrence, disease remission, new disease diagnosis and pain status including pain medication
Characterize the treatment decision as reported by the treating physician | 30 days
  Characterize the treatment decision per data provided by the treating physician (within the study database) including the rationale given for the treatment decision (e.g., age of the patient or co-morbidity); number of treatment decisions, e.g., for surgical therapy (open surgery or minimal-invasive therapy), watchful waiting, or treatment with medication will be described; descriptive analysis will be performed

SECONDARY OUTCOMES:
Investigate the impact of patient characteristics on surgery | 30 days
  Descriptive analysis of patient characteristics such as age on surgery (e.g., duration of surgery, instrument usage)
Investigate the impact of patient characteristics on clinical outcome | 30 days
  Descriptive analysis of patient characteristics such as age on clinical outcome (e.g., re-operation)
Investigate the impact of patient characteristics on complications | 30 days
  Descriptive analysis of patient characteristics such as age on complication (number of complications reported during and after the surgery)
Describe the impact from surgery to the patient's quality of life and function | 12 months
  Describe the impact from surgery to the patient's quality of life and function by comparing the baseline quality of life and functional status with the post-operative status (post-operative day 1-3, 30 days, 90 days, 6 months and 12 months)
Describe the number of Intuitive instruments used per procedure and patient characteristics | 30 days
  Describe the number of Intuitive instruments used per procedure and patient characteristics; descriptive analysis will be performed on the number of instruments used per specific procedure and patient
Describe the number of disease recurrence and re-operation at final patient follow-up | 12 months
  Describe the number disease recurrence and re-operation at final patient follow-up; descriptive analysis will be performed
Describe the number of conversion per procedure and patient characteristics | 30 days
  Describe the number conversion per procedure and patient characteristics; descriptive analysis will be performed
Describe the impact of surgeon experience on surgical times (duration of surgery per treating surgeon) | 30 days
  Describe the impact of surgeon experience on surgical times, descriptive analysis will be performed on the surgical times (duration of surgery) per treating surgeon
Describe the impact of surgeon experience on clinical outcome (number of clinical outcomes per treating surgeon) | 30 days
  Describe the impact of surgeon experience on clinical outcome; descriptive analysis will be performed, e.g., on number of re-operation or re-hospitalization per treating surgeon
Describe the impact of surgeon experience on complications (number of events per surgeon) | 30 days
  Describe the impact of surgeon experience on complications; descriptive analysis will be performed on number of adverse events per treating surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Ingolf Juhasz-Böss, Prof. Dr., Principal Investigator — Universitätsklinikum Freiburg
Locations (15):
- Germany (15):
  - Albertinen Krankenhaus Hamburg, Hamburg, Hamburg
  - St. Josefs-Hospital Wiesbaden, Wiesbaden, Hesse
  - Charité - Universitätsmedizin Berlin - Klinik für Gynäkologie, Berlin
  - Augusta-Kranken-Anstalt Bochum, Bochum
  - Sana Kliniken Coburg, Coburg
  - St. Elisabeth-Krankenhaus Köln-Hohenlind, Cologne
  - Universitätsklinikum Essen, Essen
  - Agaplesion Markus Krankenhaus Frankfurt am Main, Frankfurt am Main
  - Universitätsklinikum Freiburg - Klinik für Frauenheilkunde, Freiburg im Breisgau
  - Universitätsmedizin Greifswald, Greifswald
  - St. Ansgar Krankenhaus Höxter, Höxter
  - Universitätsklinikum Kiel, Kiel
  - Klinikum Nürnberg Nord / Klinik für Frauenheilkunde, Nuremberg
  - Helios Kliniken Schwerin, Schwerin
  - Universitätsklinikum Tübingen - Frauenklinik, Tübingen

IPD SHARING:
Plan to Share IPD: No